CLINICAL TRIAL: NCT05220566
Title: Impact of the 'Reserved Therapeutic Space' Nursing Intervention on Patient Health Outcomes: an Intervention Study in Acute Mental Health Units in Spain
Brief Title: Impact of the 'Reserved Therapeutic Space' Nursing Intervention: an Intervention Study in Acute Mental Health Units
Acronym: RTSMHNursing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Campus docent Sant Joan de Déu-Universitat de Barcelona (Other); Hospital Universitario Fundación Alcorcón (Other); Hospital Regional de Malaga (Other); Hospital Gil Casares de Santiago de Compostela (Unknown); Hospital Universitario Infanta Leonor (Other); Hospital Virgen de los Lirios de Alcoi (Unknown); Hospital Universitari de Bellvitge (Other); Hospital de Galdakao (Other); Hospital de Mataró (Other); Hospital del Mar (Other); Complejo Hospitalario Universitario de Vigo (Other); Hospital Universitario San Juan de Alicante (Other); Instituto de Salud Carlos III (Other Government); Colegio Oficial de Enfermeras y Enfermeros de Barcelona (Unknown); Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Principal Investigator, Antonio R. Moreno Poyato, PhD, Professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021/9835
Record Dates: First submitted 2021-12-16; First posted 2022-02-02 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Nurse-Patient Relations; Psychiatric Hospitalization
Keywords: Nurse-Patient therapeutic relationship; Quality of psychiatric care; Mental health nursing; Acute psychiatric care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'Reserved Therapeutic Space' (Experimental): Participants will receive 'Reserved Therapeutic Space' Nursing Intervention
  Interventions: Behavioral: Reserved Therapeutic Space
- Control (No Intervention): Participants will receive usual care

INTERVENTIONS:
Behavioral: Reserved Therapeutic Space — The main objective of the 'Reserved Therapeutic Space' intervention is to enhance the therapeutic bond of trust, to enable the agreement of objectives and interventions in a shared manner in relation to their recovery process in the unit. The intervention is carried out through individual meetings between the nurse and the patient in a comfortable and intimate space, where there are no interruptions and which is also chosen by the person who is hospitalized. The content of the spaces must be constructed individually according to the patients' concerns at each moment of the process.
  Arms: 'Reserved Therapeutic Space'

SUMMARY:
Aims:

To evaluate the effectiveness of the "Reserved Therapeutic Space" intervention for improving the nurse-patient therapeutic relationship in acute mental health units in Spain, as well as its impact in terms of quality of care and patients' perceptions of coercion.

Design:

Multicenter intervention study with control group.

Methods:

The study will be carried out in 12 mental health units in Spain. Given the conditions of evaluation in real clinical practice, paired randomization will be performed to assign centers to intervention and control groups. The "Reserved Therapeutic Space" intervention to be tested has been co-designed and validated by both nurses and patients. The quality of the therapeutic relationship, the care received, and perceived coercion among patients will be assessed at baseline and at discharge using instruments validated in our context. An estimated 131 patients per group are expected to participate. Funding was granted in July 2021 by the Institute of Health Carlos III (PI21/00605, Ministry of Science and Innovation) and in October 2021 by the College of Nurses of Barcelona (PR-487/2021). The proposal was approved by all the Research Ethics Committees of participating centers.

Discussion:

This study is expected to demonstrate the effectiveness of a specific nursing intervention on patient health outcomes including the level of the therapeutic relationship, the quality of care, the level of coercion and other specific indicators for acute mental health units.

Impact:

This project will lead to changes in clinical practice, transforming the current models of organization and care management in mental health hospitalization units, promoting the quality of the therapeutic relationship and, ultimately, the quality of person-centered care.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized in mental health inpatient units who voluntarily consent to participate in the study

Exclusion Criteria:

* Adults hospitalized in mental health inpatient units who present a language barrier, mechanical restraint, contraindication by the clinical referent, cognitive impairment, or intellectual disability at the time of recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Nurse-patient therapeutic alliance at discharge assessed by WAI-Short patient version | At baseline and at discharge from the inpatient unit (an average of 16 days)
  The Working Alliance Inventory Short Questionnaire (WAI-S), patient version. This is an instrument for measuring the working alliance, and therefore, the therapeutic relationship between professional and patient (Horvath & Greenberg, 1989). Scores range from 12-84 with higher scores indicating greater levels of therapeutic alliance.

SECONDARY OUTCOMES:
Change from baseline Quality in Psychiatric Care at discharge assessed by QPC | At baseline and at discharge from the inpatient unit (an average of 16 days)
  The Quality in Psychiatric Care scale (QPC: Schröder et al., 2007) assesses the quality of care and is the best suited to evaluate the quality of care in psychiatric units. Scores range from 30-120 with higher scores indicating greater levels of quality in psychiatric care.
Experience of coercion assessed by CES-18 | At discharge from the inpatient unit (an average of 16 days)
  The Coercion Experience Scale (CES-18: Bergk et al., 2010). This scale assesses the subjective experience of coercion during psychiatric hospitalization. Scores range from 18-90 with higher scores indicating greater levels of coercion experience.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Gil Casares, Santiago de Compostela, A Coruña
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Regional, Málaga
  - Hospital Clinic Universitari de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El-Abidi K, Moreno-Poyato AR, Canabate-Ros M, Garcia-Sanchez JA, Lluch-Canut MT, Munoz-Ruoco E, Perez-Moreno JJ, Pita-De-La-Vega J, Puig-Llobet M, Rubia-Ruiz G, Santos-Pariente C, Lopez AMR, Golmar LJ, Lopez CE, Roldan-Merino JF. The therapeutic relationship from the perspective of patients and nurses in the first days of admission: A cross-sectional study in acute mental health units. Int J Ment Health Nurs. 2024 Feb;33(1):134-142. doi: 10.1111/inm.13227. Epub 2023 Sep 24. PMID 37743558
- [Result] Moreno-Poyato AR, El Abidi K, Lluch-Canut T, Canabate-Ros M, Puig-Llobet M, Roldan-Merino JF. Impact of the 'reserved therapeutic space' nursing intervention on patient health outcomes: An intervention study in acute mental health units. Nurs Open. 2023 Aug;10(8):5749-5757. doi: 10.1002/nop2.1750. Epub 2023 Apr 21. PMID 37084278